CLINICAL TRIAL: NCT07274436
Title: The Clinical Value of Deep Learning-Based Reconstruction Techniques in Cardiac MRI Scanning
Status: Recruiting | Type: Observational
Sponsor: Lian Yang (Other)
Responsible Party: Sponsor-Investigator, Lian Yang, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2025-0804
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scanning using AI-based cardiac MRI sequences
- scanning using non-AI cardiac MRI sequences

SUMMARY:
By enrolling patients who underwent cardiac MR(Magnetic Resonance) examinations at our center and using randomized allocation, the patients were divided into a study group and a control group. The study group underwent scanning using AI-based(Artificial Intelligence-based) cardiac MRI(Magnetic Resonance Imaging) sequences, while the control group was scanned using non-AI cardiac MRI sequences

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring cardiac MRI in clinical practice;
2. Patient age ≥ 18 years;
3. The patient has signed an informed consent form.

Exclusion Criteria:

1. Patients with contraindications to magnetic resonance imaging;
2. Patients who failed to complete the MRI examination or whose image quality was inadequate for diagnostic requirements;
3. Other circumstances deemed by clinical trial personnel as unsuitable for participation in this trial;
4. Subjects or their legal guardians voluntarily requesting to withdraw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring cardiac MRI in clinical practice
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | immediately after procedure
  Patient satisfaction will be evaluated using a Likert scale with the following scoring criteria:5 - Very Satisfied;4 - Satisfied;3 - Neutral;2 - Dissatisfied;1 - Very Dissatisfied

SECONDARY OUTCOMES:
total scan time | During procedure
objective image measurements (signal-to-noise ratio) | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China